CLINICAL TRIAL: NCT00361322
Title: Topical Clindamycin Salicylic Acid Preparation for the Treatment of Acne Vulgaris
Brief Title: Efficacy and Safety of a Preparation Containing an Antibiotic and Anti-Inflammatory Agent in Acne Vulgaris
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLSA-HMO-CTIL
Record Dates: First submitted 2006-08-06; First posted 2006-08-08 (Estimated); Last update posted 2006-08-08 (Estimated); Status verified 2006-08

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — clindamycin phosphate; Salicylic Acid

INTERVENTIONS:
Drug: clindamycin phosphate
Drug: salicylic acid

SUMMARY:
The concept behind our study was to combine an effect of antibiotic and anti-inflammatory agents for a more efficient acne therapy directed at the factors involved in the pathophysiology of the disease. For this purpose we evaluated a combination of clindamycin phosphate and salicylic acid in a non-irritating carrier.

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate acne vulgaris;
* at least 5 lesions on the face;
* a one-month wash-out period was established for any topical or systemic drug use for treatment of acne vulgaris.

Exclusion Criteria:

* acne that was primarily truncal, nodular, or due to secondary causes/internal disease;
* pregnancy, breastfeeding, or intention to become pregnant;
* another dermatological disease of the face;
* significant systemic disease;
* any drug/alcohol addiction;
* interacting medication;
* known hypersensitivity to study medications;
* history of chronic disease treated with medications which might affect acne condition and treatment outcome (e.g. corticosteroids, lithium, isoniazid, anti-androgens, phenytoin, phenobarbital) in the preceding month

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Enrollment: 40
Dates: Start 2005-04; Study Completion 2006-01

PRIMARY OUTCOMES:
Lesions count at the baseline (week 0)
Lesions count at the end of study (week 8)

CONTACTS AND LOCATIONS:
Overall Officials: Vera Leibovici, MD, Principal Investigator — Hadassah Medical Organization; Arie Ingber, MD, Prof, Principal Investigator — Hadassah Medical Organization; Elka Touitou, PhD, Prof, Principal Investigator — The Hebrew University of Jerusalem, Jerusalem, Israel
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel